CLINICAL TRIAL: NCT05063487
Title: Evaluating the Impact of HIV-1 Recent Infection Testing on Incremental HIV Testing Yield and Adverse Events Linked to Return of Recent Infection Testing Results in Rwanda
Brief Title: Evaluation of HIV-1 Recent Infection Testing in Rwanda
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Ministry of Health, Rwanda (Other Government)
Responsible Party: Principal Investigator, Suzue Saito, Associate Research Scientist in ICAP, Columbia University
Other Study IDs: AAAT5637; GG014256-18 (Other Grant/Funding Number: CDC)
Record Dates: First submitted 2021-09-13; First posted 2021-10-01 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: HIV Infections
Keywords: HIV Infections; HIV-1; Rapid Test for Recent Infection; RTRI; recent infection; newly diagnosed people living with HIV
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Recent HIV Infection: Persons ≥15 years of age who are newly-diagnosed with HIV, consent to participate in case-based surveillance and recency testing and test recent on the rapid test for recent infection (RTRI).
  Interventions: Other: Return of recent classification
- Long-Term HIV Infection: Persons ≥15 years of age who are newly-diagnosed with HIV, consent to participate in case-based surveillance and recency testing and test long-term on the rapid test for recent infection (RTRI).
  Interventions: Other: Return of long-term classification

INTERVENTIONS:
Other: Return of recent classification — As part of routine HIV case-based surveillance in Rwanda, blood samples are collected for recency testing on the Rapid Test for Recent Infection (RTRI) assay and viral load testing for all newly diagnosed people living with HIV. Results of a recent classification (i.e., having acquired an HIV infection within the last year) will be returned to study participants during a scheduled 1-month visit following initial HIV diagnosis.
  Groups: Recent HIV Infection
Other: Return of long-term classification — As part of routine HIV case-based surveillance in Rwanda, blood samples are collected for recency testing on the Rapid Test for Recent Infection (RTRI) assay and viral load testing for all newly diagnosed people living with HIV. Results of a long-term classification (i.e., having acquired an HIV infection more than one year ago) will be returned to study participants during the scheduled 1-month visit following initial HIV diagnosis.
  Groups: Long-Term HIV Infection

SUMMARY:
The study is a longitudinal, observational cohort study of people who are newly-diagnosed with HIV who consent to recency testing and participate in index testing services, and their disclosed contacts.

The study will evaluate the impact of recency testing on HIV positive yield of index testing among the contacts of newly diagnosed people living with HIV and the incidence of adverse events or social harm as a result of returning recency results among newly diagnosed people living with HIV.

DETAILED DESCRIPTION:
The rapid test for recent HIV infection (RTRI) assay can distinguish between people who are recently-infected and those who are long-term HIV cases. This may help guide efforts to identify ongoing HIV transmission and direct prevention or treatment efforts. But, more research is needed on the impact of RTRI on the number of HIV+ individuals that can be identified through testing. Furthermore, not much is known about the impact that returning RTRI results may have on the occurrence of intimate partner violence.

A primary objective of this study is to compare the HIV testing yield among contacts of people newly diagnosed with HIV by recency testing result. The investigators will abstract routinely collected data from participant medical records and registers. In addition, a second primary objective of this study is to assess the incidence of intimate partner violence associated with the return of recency testing results among those classified as testing recent versus long-term. Index study participants newly diagnosed with HIV will be interviewed at the initial enrollment visit following HIV diagnosis and during follow-up visits at 1, 2, and 6-months using a health-related quality of life instrument and intimate partner violence questionnaire. Participants will be recruited from 60 high-volume facilities across all provinces in Rwanda during the evaluation period.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥15 years
* Be newly diagnosed with HIV
* Ability to speak and understand English or Kinyarwanda
* Consented to be part of both case-based surveillance (CBS) (which includes PNS) and recency surveillance under the separate, approved CBS protocol.
* Give voluntary written informed consent for data collection via semi-structured interview and survey instruments
* Give voluntary written informed consent for use of routinely collected data
* Be female if they are received at the facility at the same time as their partner (for intimate partner violence objective only).

Exclusion Criteria:

* Opt out or do not consent, or are unable to consent to participate in semi-structured interviews and completion of survey instruments
* Have a history of testing HIV positive (i.e., not newly diagnosed with HIV)
* Report antiretroviral drug (ARV) use for HIV management at any point during the HIV testing service (HTS) visit

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population are persons ≥15 years of age who are newly diagnosed with HIV during HIV testing services (i.e., a previously undiagnosed HIV case) and who provide informed consent for their blood to be tested for recent HIV infection.
Sampling Method: Non-Probability Sample
Enrollment: 1588 (Actual)
Dates: Start 2021-07-29 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
The HIV positive yield of index testing among the contacts of people newly diagnosed with HIV that test recent versus long-term. | From baseline to 6 months after initial diagnosis
  We will compare the number of HIV positive contacts that are linked to HIV recent vs. long-term index cases newly diagnosed with HIV.
The incidence of intimate partner violence associated with the return of recency testing results among people newly diagnosed with HIV that test recent versus long-term | From baseline to 6 months after initial HIV diagnosis
  We will compare the incremental change in intimate partner violence resulting from the return of recency testing results between 2 and 6 months, adjusting for baseline and 1 month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Suzue Saito, PhD, Principal Investigator — Columbia University; Gallican Rwibasira, MD, Principal Investigator — Rwanda Biomedical Centre
Locations (1):
- Rwanda Biomedical Centre, Ministry of Health, Kigali, Rwanda

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data (with removal of personally identifiable data) will be made available concurrently with the release of the final report to a dedicated website where requests for data can be submitted.
Time Frame: Individual Participant Data will be made publicly available approximately six months after the final data set is made available to investigators.
Access Criteria: A de-identified dataset will be made available publicly to a dedicated website. Requestors of Individual Participant Data will submit requests and data will be released to all bona fide. requesting institutions and individuals.